CLINICAL TRIAL: NCT00866047
Title: A Phase 2 Study of SGN-35 in Treatment of Patients With Relapsed or Refractory Systemic Anaplastic Large Cell Lymphoma (ALCL)
Brief Title: A Phase 2 Open Label Trial of Brentuximab Vedotin (SGN-35) for Systemic Anaplastic Large Cell Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Seagen Inc. (Industry)
Collaborators: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SG035-0004; 2008-006035-12 (EudraCT Number)
Record Dates: First submitted 2009-03-19; First posted 2009-03-20 (Estimated); Results first posted 2011-10-26 (Estimated); Last update posted 2017-03-22 (Actual); Status verified 2016-12

CONDITIONS: Lymphoma, Large-Cell, Anaplastic; Lymphoma, Non-Hodgkin
Keywords: Antigens, CD30; Antibody-Drug Conjugate; Antibodies, Monoclonal; Lymphoma, Non-Hodgkin; Lymphoma, Large-Cell, Anaplastic; monomethyl auristatin E; Drug Therapy; Immunotherapy; Hematologic Diseases; Lymphoma
MeSH Terms: conditions — Lymphoma, Large-Cell, Anaplastic; Lymphoma, Non-Hodgkin; Hematologic Diseases; Lymphoma | interventions — Brentuximab Vedotin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Brentuximab vedotin (Experimental): Brentuximab vedotin 1.8 mg/kg every 3 weeks by intravenous (IV) infusion
  Interventions: Drug: brentuximab vedotin

INTERVENTIONS:
Drug: brentuximab vedotin — 1.8 mg/kg every 3 weeks by IV infusion
  Other Names: SGN-35; ADCETRIS

SUMMARY:
This is a single-arm, open-label, multicenter, clinical trial to evaluate the efficacy and safety of brentuximab vedotin (SGN-35) as a single agent in patients with relapsed or refractory ALCL.

ELIGIBILITY:
Inclusion Criteria:

* Patients with relapsed or refractory systemic ALCL who have previously received front line chemotherapy.
* Documented anaplastic lymphoma kinase (ALK) status.
* Histologically-confirmed CD30-positive disease; tissue from the most recent post diagnostic biopsy of relapsed/refractory disease must be available for confirmation of CD30 expression via slides or tumor block.
* Fluorodeoxyglucose-avid and measurable disease of at least 1.5 cm as documented by both positron emission tomography and spiral computed tomography.
* Received any previous autologous stem cell transplant at least 12 weeks (3 months) prior.
* At US sites, patients greater than or equal to 12 years of age may be enrolled. At non-US sites, patients must be greater than or equal to 18 years of age.

Exclusion Criteria:

* Previous treatment with brentuximab vedotin.
* Previously received an allogeneic transplant.
* Patients with current diagnosis of primary cutaneous ALCL (patients who have transformed to systemic ALCL are eligible).
* Known cerebral/meningeal disease.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2009-03; Primary Completion 2010-08 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dana Kennedy, PharmD, Study Director — Seagen Inc.
Locations (22):
- United States (15):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Stanford University Medical Center, Palo Alto, California
  - Rocky Mountain Cancer Centers, Denver, Colorado
  - University of Miami Sylvester Comprehensive Cancer Center, Miami, Florida
  - Northwestern University, Chicago, Illinois
  - Karmanos Cancer Institute / Wayne State University, Detroit, Michigan
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Weill Cornell Medical College, New York, New York
  - Nationwide Children's Hospital, Columbus, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - Baylor Sammons Cancer Center / Texas Oncology, Dallas, Texas
  - MD Anderson Cancer Center / University of Texas, Houston, Texas
  - University of Washington, Seattle, Washington
- UZ Gasthuisberg, Leuven, Belgium
- Canada (2):
  - B.C Cancer Agency, Vancouver, British Columbia
  - Princess Margaret Hospital, Toronto, Ontario
- France (3):
  - Institut Paoli Calmettes, Marseille
  - Hospital Saint Louis, Paris
  - Centre Henri Becquerel, Rouen
- Christie Hospital NHS, Manchester, United Kingdom

REFERENCES:
- [Result] Pro B, Advani R, Brice P, Bartlett NL, Rosenblatt JD, Illidge T, Matous J, Ramchandren R, Fanale M, Connors JM, Yang Y, Sievers EL, Kennedy DA, Shustov A. Brentuximab vedotin (SGN-35) in patients with relapsed or refractory systemic anaplastic large-cell lymphoma: results of a phase II study. J Clin Oncol. 2012 Jun 20;30(18):2190-6. doi: 10.1200/JCO.2011.38.0402. Epub 2012 May 21. PMID 22614995
- [Derived] Pro B, Advani R, Brice P, Bartlett NL, Rosenblatt JD, Illidge T, Matous J, Ramchandren R, Fanale M, Connors JM, Fenton K, Huebner D, Pinelli JM, Kennedy DA, Shustov A. Five-year results of brentuximab vedotin in patients with relapsed or refractory systemic anaplastic large cell lymphoma. Blood. 2017 Dec 21;130(25):2709-2717. doi: 10.1182/blood-2017-05-780049. Epub 2017 Oct 3. PMID 28974506

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment period: Jun 2009 - May 2010
Period: Treatment Period
Arm/Group | Brentuximab Vedotin
Started | 58
Completed | 10 (Number who completed 16 cycles of treatment)
Not Completed | 48
Not completed — Progressive disease | 13
Not completed — Adverse Event | 16
Not completed — Physician Decision | 14
Not completed — Withdrawal by Subject | 5
Period: Follow-up Period
Arm/Group | Brentuximab Vedotin
Started | 58 (All participants were to be followed after treatment)
Completed | 53 (Completed survival follow-up due to death [25] or study completion [28])
Not Completed | 5
Not completed — Lost to Follow-up | 5

BASELINE CHARACTERISTICS:
Groups:
- Brentuximab Vedotin: Brentuximab vedotin 1.8 mg/kg every 3 weeks by IV infusion
Arm/Group | Brentuximab Vedotin
Number analyzed (Participants) | 58
Age, Customized [Median (Full Range); unit: years] | 52.0 [14 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 33
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 7
  White | 48
  More than one race | 0
  Unknown or Not Reported | 2
Eastern Cooperative Oncology Group Performance Status [Number; unit: participants] — 0 = Normal activity
  1. = Symptoms but ambulatory
  2. = In bed <50% of the time
  3. = In bed >50% of the time
  4. = 100% bedridden
  5. = Dead
  participants
    0 | 19
    1 | 38
    2 | 1
    3-5 | 0
ALK Status [Number; unit: participants] — Immunophenotype status with respect to anaplastic lymphoma kinase (ALK) protein
  participants
    Positive | 16
    Negative | 42

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate by Independent Review Group
Description: Percentage of participants who achieved a best response of complete remission (CR, disappearance of all evidence of disease) or partial remission (PR, regression of greater than or equal to 50% of measurable disease and no new sites) per Cheson 2007 Revised Response Criteria for Malignant Lymphoma.
Time Frame: up to 12 months
Population: Intention to treat
Measure: Number (95% Confidence Interval); unit: percent of participants
Arm/Group | Brentuximab Vedotin
Number analyzed (Participants) | 58
percent of participants | 86 [74.6 to 93.9]

2. Secondary Outcome: Complete Remission Rate by Independent Review Group
Description: Percentage of participants who achieved a best response of CR (disappearance of all evidence of disease) per Cheson 2007 Revised Response Criteria for Malignant Lymphoma.
Time Frame: up to 12 months
Population: Intention to treat
Measure: Number (95% Confidence Interval); unit: percent of participants
Arm/Group | Brentuximab Vedotin
Number analyzed (Participants) | 58
percent of participants | 59 [44.9 to 71.4]

3. Secondary Outcome: Duration of Objective Response by Kaplan-Meier Analysis
Description: Duration of objective response (CR + PR) by independent review group, defined as time of initial response until disease progression or death.
Time Frame: up to approximately 3 years
Population: Participants with objective response among the intention to treat population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Brentuximab Vedotin
Number analyzed (Participants) | 50
months | 13.2 [5.7 to 26.3]

4. Secondary Outcome: Duration of Objective Response in Participants With Complete Remission by Kaplan-Meier Analysis
Description: Duration of response from start of first objective tumor response (CR or PR) by independent review group to disease progression or death due to any cause in participants with CR.
Time Frame: up to approximately 3 years
Population: Participants with complete remission among the intention to treat population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Brentuximab Vedotin
Number analyzed (Participants) | 34
months | 26.3 [13.2 to NA] — Insufficient number of events to estimate upper bound

5. Secondary Outcome: Progression-free Survival by Kaplan-Meier Analysis
Description: Time from start of study treatment to disease progression per independent review group or death due to any cause.
Time Frame: up to approximately 3 years
Population: Intention to treat
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Brentuximab Vedotin
Number analyzed (Participants) | 58
months | 14.6 [6.9 to 20.6]

6. Secondary Outcome: Overall Survival
Description: Time from start of study treatment to date of death due to any cause.
Time Frame: up to approximately 7 years
Population: Intention to treat
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Brentuximab Vedotin
Number analyzed (Participants) | 58
months | NA [21.3 to NA] — Insufficient number of events to estimate median and upper bound

7. Secondary Outcome: Adverse Events by Severity, Seriousness, and Relationship to Treatment
Description: Counts of participants who had adverse events or treatment-emergent adverse events (TEAE, defined as newly occurring or worsening after first dose). Serious adverse events are reported from the time of informed consent. National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE version 3.0) were used to assess severity (1=mild, 2=moderate, 3=severe, 4=life threatening/disabling, 5=death). Relatedness to study drug was assessed by the investigator (Yes/No). Participants with multiple occurrences of an adverse event within a category are counted once within the category.
Time Frame: up to 12 months
Population: All participants who received treatment
Measure: Number; unit: participants
Arm/Group | Brentuximab Vedotin
Number analyzed (Participants) | 58
participants
  Any TEAE | 58
  TEAE related to study drug | 53
  TEAE with CTCAE severity grade >/=3 | 36
  Serious adverse event | 25
  Serious adverse event related to study drug | 11
  Discontinued treatment due to adverse event | 16

8. Secondary Outcome: Hematology Laboratory Abnormalities >/= Grade 3
Description: Counts of study participants with post-baseline hematology laboratory abnormalities of Grade 3 or greater per NCI CTCAE version 3.0. Participants with multiple occurrences of a laboratory abnormality within a category are counted once in that category.
Time Frame: up to 12 months
Population: All participants who received treatment
Measure: Number; unit: participants
Arm/Group | Brentuximab Vedotin
Number analyzed (Participants) | 58
participants
  Any >/= Grade 3 hematology laboratory abnormality | 17
  Leukocytes (low) | 3
  Lymphocytes (low) | 10
  Neutrophils (low) | 7
  Platelets (low) | 3

9. Secondary Outcome: Chemistry Laboratory Abnormalities >/= Grade 3
Description: Counts of study participants with post-baseline chemistry laboratory abnormalities of Grade 3 or greater per NCI CTCAE version 3.0. Participants with multiple occurrences of a laboratory abnormality within a category are counted once in that category.
Time Frame: up to 12 months
Population: All participants who received treatment
Measure: Number; unit: participants
Arm/Group | Brentuximab Vedotin
Number analyzed (Participants) | 58
participants
  Any >/= Grade 3 chemistry laboratory abnormality | 13
  Aspartate aminotransferase (high) | 1
  Calcium (low) | 3
  Glucose (high) | 4
  Potassium (low) | 1
  Sodium (low) | 1
  Urate (high) | 3

10. Secondary Outcome: Area Under the Curve
Description: Area under the serum concentration-time curve from time 0 to 21 days following the first dose of brentuximab vedotin
Time Frame: 3 weeks
Population: All participants who received treatment
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: day * microgram/mL
Arm/Group | Brentuximab Vedotin
Number analyzed (Participants) | 58
day * microgram/mL | 98 (69)

11. Other Pre Specified Outcome: B Symptom Resolution
Description: Percentage of participants with lymphoma-related symptoms (B symptoms: fever, night sweats, or weight loss >10%) at baseline who achieved resolution of all B symptoms at any time during the treatment period.
Time Frame: up to 12 months
Population: Participants with B symptoms at baseline
Measure: Number (95% Confidence Interval); unit: percent of participants
Arm/Group | Brentuximab Vedotin
Number analyzed (Participants) | 17
percent of participants | 82 [56.6 to 96.2]

12. Secondary Outcome: Maximum Serum Concentration
Description: Maximum serum concentration from 0 to 21 days following the first dose of brentuximab vedotin
Time Frame: 3 weeks
Population: All participants who received treatment
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram/mL
Arm/Group | Brentuximab Vedotin
Number analyzed (Participants) | 58
microgram/mL | 37 (20)

13. Secondary Outcome: Time of Maximum Serum Concentration
Description: Time of maximum serum concentration from 0 to 21 days following the first dose of brentuximab vedotin
Time Frame: 3 weeks
Population: All participants who received treatment
Measure: Median (Full Range); unit: days
Arm/Group | Brentuximab Vedotin
Number analyzed (Participants) | 58
days | 0.02 [0.02 to 0.02]

ADVERSE EVENTS:
Time Frame: Adverse events through 30 days after last dose (up to 12 months)
Arm/Group | Brentuximab Vedotin
Serious Adverse Events (participants affected / at risk) | 25/58
Other Adverse Events (participants affected / at risk) | 58/58
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Brentuximab Vedotin (N=58)
Anaemia (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 1
Acute myocardial infarction (Cardiac disorders) | 1
Arrhythmia supraventricular (Cardiac disorders) | 2
Atrial fibrillation (Cardiac disorders) | 1
Atrioventricular block complete (Cardiac disorders) | 1
Bradycardia (Cardiac disorders) | 1
Retinal vein occlusion (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Asthenia (General disorders) | 1
Generalised oedema (General disorders) | 1
Sudden death (General disorders) | 1
Cellulitis (Infections and infestations) | 1
Endocarditis staphylococcal (Infections and infestations) | 1
Gastroenteritis viral (Infections and infestations) | 1
Klebsiella bacteraemia (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Septic shock (Infections and infestations) | 2
Superinfection bacterial (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 2
Lower limb fracture (Injury, poisoning and procedural complications) | 1
Decreased appetite (Metabolism and nutrition disorders) | 1
Fluid overload (Metabolism and nutrition disorders) | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1
Tumour lysis syndrome (Metabolism and nutrition disorders) | 1
Myositis (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2
Anaplastic large cell lymphoma t- and null-cell types recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Mycosis fungoides (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Tumour flare (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Encephalopathy (Nervous system disorders) | 1
Haemorrhage intracranial (Nervous system disorders) | 1
Neuralgia (Nervous system disorders) | 1
Peripheral motor neuropathy (Nervous system disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1
Spinal cord compression (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Mental status changes (Psychiatric disorders) | 1
Hydronephrosis (Renal and urinary disorders) | 1
Renal failure (Renal and urinary disorders) | 1
Renal failure acute (Renal and urinary disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Tracheal disorder (Respiratory, thoracic and mediastinal disorders) | 1
Rash papular (Skin and subcutaneous tissue disorders) | 1
Deep vein thrombosis (Vascular disorders) | 1
Demyelinating polyneuropathy (Nervous system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Brentuximab Vedotin (N=58)
Anaemia (Blood and lymphatic system disorders) | 5
Lymphadenopathy (Blood and lymphatic system disorders) | 6
Neutropenia (Blood and lymphatic system disorders) | 11
Thrombocytopenia (Blood and lymphatic system disorders) | 8
Abdominal distension (Gastrointestinal disorders) | 3
Abdominal pain (Gastrointestinal disorders) | 5
Constipation (Gastrointestinal disorders) | 12
Diarrhoea (Gastrointestinal disorders) | 16
Dyspepsia (Gastrointestinal disorders) | 5
Nausea (Gastrointestinal disorders) | 23
Oral pain (Gastrointestinal disorders) | 5
Vomiting (Gastrointestinal disorders) | 9
Asthenia (General disorders) | 5
Chills (General disorders) | 8
Fatigue (General disorders) | 22
Oedema peripheral (General disorders) | 8
Pain (General disorders) | 6
Pyrexia (General disorders) | 20
Bronchitis (Infections and infestations) | 3
Folliculitis (Infections and infestations) | 5
Upper respiratory tract infection (Infections and infestations) | 11
Excoriation (Injury, poisoning and procedural complications) | 3
Weight decreased (Investigations) | 8
Decreased appetite (Metabolism and nutrition disorders) | 8
Dehydration (Metabolism and nutrition disorders) | 3
Hyperglycaemia (Metabolism and nutrition disorders) | 3
Hypokalaemia (Metabolism and nutrition disorders) | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 5
Back pain (Musculoskeletal and connective tissue disorders) | 5
Groin pain (Musculoskeletal and connective tissue disorders) | 5
Muscle spasms (Musculoskeletal and connective tissue disorders) | 8
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 9
Neck pain (Musculoskeletal and connective tissue disorders) | 5
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6
Tumour flare (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4
Dizziness (Nervous system disorders) | 9
Headache (Nervous system disorders) | 11
Paraesthesia (Nervous system disorders) | 5
Peripheral motor neuropathy (Nervous system disorders) | 3
Peripheral sensory neuropathy (Nervous system disorders) | 24
Anxiety (Psychiatric disorders) | 4
Confusional state (Psychiatric disorders) | 3
Depression (Psychiatric disorders) | 4
Insomnia (Psychiatric disorders) | 9
Cough (Respiratory, thoracic and mediastinal disorders) | 10
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 11
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4
Productive cough (Respiratory, thoracic and mediastinal disorders) | 3
Alopecia (Skin and subcutaneous tissue disorders) | 8
Dermatitis (Skin and subcutaneous tissue disorders) | 4
Dry skin (Skin and subcutaneous tissue disorders) | 6
Night sweats (Skin and subcutaneous tissue disorders) | 4
Pruritus (Skin and subcutaneous tissue disorders) | 11
Rash (Skin and subcutaneous tissue disorders) | 14
Rash pruritic (Skin and subcutaneous tissue disorders) | 4
Hot flush (Vascular disorders) | 3
Anaplastic large cell lymphoma t- and null-cell types recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Hypomagnesaemia (Metabolism and nutrition disorders) | 3
Nasopharyngitis (Infections and infestations) | 3
Sinusitis (Infections and infestations) | 4
Tachycardia (Cardiac disorders) | 3
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3
Haemorrhoids (Gastrointestinal disorders) | 3
Memory impairment (Nervous system disorders) | 3
Neuralgia (Nervous system disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less